CLINICAL TRIAL: NCT02348008
Title: Phase Ib and Phase II Studies of Anti-PD-1 Antibody MK-3475 in Combination With Bevacizumab for the Treatment of Metastatic Renal Cell Carcinoma: Big Ten Cancer Research Consortium GU14-003
Brief Title: Phase Ib and Phase II Studies of MK-3475 in Combination + for Renal Cell Carcinoma:
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arkadiusz Z. Dudek, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Big Ten Cancer Research Consortium (Other)
Responsible Party: Sponsor-Investigator, Arkadiusz Z. Dudek, MD, Sponsor-Investigator, Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC GU14-003
Record Dates: First submitted 2015-01-16; First posted 2015-01-28 (Estimated); Results first posted 2020-07-31 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-08

CONDITIONS: Clear Cell Renal Carcinoma
Keywords: MK-3475; Pembrolizumab; Bevacizumab
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pembrolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A - Phase 1b Dose Escalation Cohort (Experimental): Cohort 1 will consist of 3-6 patients who will receive MK-3475 200mg and bevacizumab 10mg on day 1 of the 21-day cycle. The drugs are administered 15-30 minutes apart in separate intravenous infusions.
  Cohort 2 will consist of 3-9 patients who will receive MK-3475 200mg and bevacizumab 15mg on day 1 of the 21-day cycle. The drugs are administered 15-30 minutes apart in separate intravenous infusions.
  If none of the 3 subjects experience a dose limiting toxicity (DLT) during the first cycle of therapy, an additional 3 subjects will be enrolled at dose level 2. If all three subjects in dose level 2 complete the first cycle of therapy without DLT, 3 more subjects will be enrolled to ensure only 0-1 of 6 subjects have a DLT. There will be no further escalation beyond dose level 2.
  Interventions: Drug: MK-3475; Drug: Bevacizumab
- Arm B - Phase II Investigational Treatment (Other): The maximum safe dose of MK-3475 in combination bevacizumab (as determined in the phase 1b cohort) will be given on day 1 of each 21 day cycle.
  Interventions: Drug: MK-3475; Drug: Bevacizumab

INTERVENTIONS:
Drug: MK-3475 — Arm A: Phase 1b Cohort 1: 200mg IV; Arm A: Phase 1b Cohort 2: 200mg IV
  Other Names: Pembrolizumab
  Arms: Arm A - Phase 1b Dose Escalation Cohort
Drug: Bevacizumab — Arm A: Phase 1b Cohort 1: 10mg IV; Arm A: Phase 1b Cohort 2: 15mg IV
  Other Names: Avastin
  Arms: Arm A - Phase 1b Dose Escalation Cohort
Drug: MK-3475 — Arm B: Phase II Treatment: 200mg IV
  Other Names: Pembrolizumab
  Arms: Arm B - Phase II Investigational Treatment
Drug: Bevacizumab — Arm B: Phase II Treatment: administered at the maximum safe dose of 10mg or 15mg as established in the Phase 1b dose escalation cohort study.
  Other Names: Avastin
  Arms: Arm B - Phase II Investigational Treatment

SUMMARY:
This is an open label, multi-institutional, single arm study of dose escalation phase Ib cohort, followed by a phase II cohort of anti-PD-1 antibody MK-3475 in combination with bevacizumab. No randomization or blinding is involved.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

The phase Ib dose escalation study will evaluate MK-3475 in combination with bevacizumab in subjects with metastatic clear cell renal carcinoma after failure of at least one systemic therapy for metastatic disease. The phase II trial will determine the activity of the combination of MK-3475 and bevacizumab in first line therapy for subjects with metastatic clear cell renal carcinoma.

PHASE Ib DOSE ESCALATION INVESTIGATIONAL TREATMENT:

Cohort 1 will consist of 3-6 patients who will receive MK-3475 200mg and bevacizumab 10mg on day 1 of the 21-day cycle. The drugs are administered 15-30 minutes apart in separate intravenous infusions.

Cohort 2 will consist of 3-9 patients who will receive MK-3475 200mg and bevacizumab 15mg on day 1 of the 21-day cycle. The drugs are administered 15-30 minutes apart in separate intravenous infusions.

If none of the 3 subjects experience a dose limiting toxicity (DLT) during the first cycle of therapy, an additional 3 subjects will be enrolled at dose level 2. If all three subjects in dose level 2 complete the first cycle of therapy without DLT, 3 more subjects will be enrolled to ensure only 0-1 of 6 subjects have a DLT. There will be no further escalation beyond dose level 2.

PHASE II INVESTIGATIONAL TREATMENT:

The maximum safe dose of MK-3475 in combination bevacizumab (as determined in the phase 1b cohort) will be given on day 1 of each 21 day cycle. Treatment will continue until disease progression, unacceptable toxicity, subject refusal, or subject death either from progression of disease, the therapy itself, or from other causes. Subjects who voluntarily stop the study, have progressive disease, or unacceptable toxicities will be followed for a total of 24 months.

Karnofsky Performance Status (KPS) ≥ 70% within 28 days prior to registration for protocol therapy.

Life Expectancy: 6 months or greater

The following baseline labs must be completed within 28 days prior to registration for protocol therapy:

Hematopoietic:

* Absolute neutrophil count (ANC) ≥ 1.5 × 10 9/L
* Platelets ≥ 100 × 10 9/L
* Hemoglobin (Hgb) ≥ 9.0 g/dL

Renal:

* Serum creatinine ≤ 1.5 × upper limit of normal (ULN)
* OR, if serum creatinine > 1.5 × ULN, estimated glomerular filtration rate (eGFR) ≥ 40 mL/min

Hepatic:

* Total serum bilirubin ≤ 1.5 × ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN
* OR, AST and ALT ≤ 5 × ULN if liver function abnormalities are due to underlying malignancy

Coagulation:

* INR < 1.5 × ULN
* OR for subjects receiving warfarin or LMWH, the subjects must, in the investigator's opinion, be clinically stable with no evidence of active bleeding while receiving anticoagulant therapy. The INR for these subjects may exceed 1.5 × ULN if that is the goal of anticoagulant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age at time of consent.
* Phase Ib dose escalation cohort study: subjects with histologically assessed metastatic clear cell RCC (defined as more than 50% clear cell component) after failure of at least one systemic therapy for metastatic disease (including, but not limited to prior therapy with interleukin 2, interferon, bevacizumab, VEGF TKI, and mTOR) for metastatic disease. NOTE: A biopsy to prove metastatic disease is not required.
* Phase II study: subjects with treatment-naïve histologically assessed metastatic clear cell RCC (defined as more than 50% clear cell component) and who are candidates for standard first-line therapy. NOTE: A biopsy to prove metastatic disease is not required.
* Measurable disease, defined as at least 1 tumor that fulfills the criteria for a target lesion according to RECIST 1.1, and obtained by imaging within 28 days prior to registration for protocol therapy.
* Karnofsky Performance Status ≥ 70% within 28 days prior to registration for protocol therapy.
* Life expectancy of 6 months or greater as determined by the treating physician.
* Adequate hepatic function within 28 days prior to registration for protocol therapy defined as meeting all of the following criteria:

  * total bilirubin ≤ 1.5 × upper limit of normal (ULN) OR direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 x ULN
  * and aspartate aminotransferase (AST) ≤ 2.5 × ULN or ≤ 5 × ULN for subjects with known hepatic metastases
  * and alanine aminotransferase (ALT) ≤ 2.5 × ULN or ≤ 5 × ULN for subjects with known hepatic metastases
* Adequate renal function within 28 days prior to registration for protocol therapy defined by either of the following criteria:

  * serum creatinine ≤ 3 mg/dL
  * OR if serum creatinine > 3 mg/dL, estimated glomerular filtration rate (GFR) ≥ 20 mL/min
* Adequate hematologic function within 28 days prior to registration for protocol therapy defined as meeting all of the following criteria:

  * hemoglobin ≥ 9 g/dL
  * and absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L
  * and platelet count ≥ 100 × 10^9/L
* Adequate coagulation functioning within 28 days prior to registration for protocol therapy defined by either of the following criteria:

  * INR < 1.5 × ULN
  * OR for subjects receiving warfarin or LMWH, the subjects must, in the investigator's opinion, be clinically stable with no evidence of active bleeding while receiving anticoagulant therapy. The INR for these subjects may exceed 1.5 × ULN if that is the goal of anticoagulant therapy.
* Provided written informed consent and HIPAA authorization for release of personal health information, approved by an Institutional Review Board/Independent Ethics Committee (IRB/IEC).
* Women of childbearing potential (WOCP) must not be pregnant or breast-feeding. A negative serum or urine pregnancy test is required within 72 hours of study registration. If the urine test cannot be confirmed as negative, a serum pregnancy test will be required.
* Women of childbearing potential (WOCP) must be willing to use two effective methods of birth control such as an oral, implantable, injectable, or transdermal hormonal contraceptive, an intrauterine device (IUD), use of a double barrier method (condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream), or total abstinence for the course of the study until 120 days after the last dose of study drug.
* Men who are not surgically sterile (vasectomy) must agree to use an acceptable method of contraception. Male subjects with female sexual partners who are pregnant, possibly pregnant, or who could become pregnant during the study must agree to use condoms from the first dose of study drug through at least 120 days after the last dose of study drug. Total abstinence for the same study period is an acceptable alternative.
* Availability of tissue if applicable (from the primary tumor or metastases) for correlative studies.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Phase Ib: Received prior monoclonal antibody therapy other than bevacizumab within 4 weeks of study registration or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events of such agents administered more than 4 weeks earlier.
* Phase II: has had prior therapy for metastatic renal cell carcinoma.
* Surgery within 4 weeks prior to study treatment except for minor procedures: NOTES: Hepatic biliary stent placement is allowed. Subject must have adequately recovered from the toxicity and/or complications of major surgery prior to study registration, as determined by the treating physician.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with neurological symptoms must undergo a head CT scan or brain MRI to exclude brain metastasis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to study registration. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
* Previously received an organ or allogeneic progenitor/stem cell transplant.
* Received a live vaccine within 30 days prior to the first dose of trial treatment: Examples of live vaccines include, but are not limited to: measles, mumps, rubella, chicken pox, yellow fever, rabies, BCG, and typhoid (oral) vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. Flu-Mist®) are live attenuated vaccines and are not allowed.
* History of blood clots, pulmonary embolism, or deep vein thrombosis unless controlled by anticoagulant treatment.
* Known history of human immunodeficiency virus [(HIV) HIV 1/2 antibodies].
* Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to study registration.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).

NOTE: Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.

* Received prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study registration or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events from previously administered agents. NOTE: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and can still be considered for the study.
* Any clinically significant infection defined as any acute viral, bacterial, or fungal infection that requires specific treatment. NOTE: Anti-infective treatment must be completed ≥ 7 days prior to study registration.
* Evidence of interstitial lung disease, history of (non-infectious) pneumonitis that required steroids, or current pneumonitis.
* Known history of active tuberculosis.
* Any other severe, uncontrolled medical condition, including uncontrolled diabetes mellitus or unstable congestive heart failure.
* Known allergy to pembrolizumab or any of its excipients.
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies.
* Any condition that, in the opinion of the treating physician, would exclude the subject from receiving bevacizumab. Examples may include but are not limited to:

  * Hemoptysis (defined as > ½ teaspoon of blood)
  * Pre-existing bleeding diathesis, coagulopathy or hemorrhage
  * Myocardial infarction or cerebrovascular accident within 6 months prior to study registration
  * Any drugs or supplements that interfere with blood clotting can raise the risk of bleeding during treatment with bevacizumab. These drugs include vitamin E, non-steroidal anti-inflammatory drugs (NSAIDs) such as aspirin, ibuprofen (Advil, Motrin), and naproxen (Aleve, Naprosyn), warfarin (Coumadin), ticlopidine (Ticlid), and clopidogrel (Plavix).These agents should be used with caution.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for enrollment in this study.
* Presence of any non-healing wound, fracture, or ulcer within 28 days prior to study registration.
* Any condition that, in the opinion of the investigator, might jeopardize the safety of the subject or interfere with protocol compliance.
* Any mental or medical condition that prevents the subject from giving informed consent or participating in the trial.
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, Gleason ≤ grade 7 prostate cancers, or other cancer for which the subject has been disease-free for at least 5 years.
* Received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Treatment with any investigational agent within 28 days prior to registration for protocol therapy and the subject must have recovered from the acute toxic effects of the regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arkadiusz Z Dudek, M.D., Ph.D., Study Chair — Big Ten Cancer Research Consortium
Locations (9):
- United States (9):
  - Northwestern University, Robert H. Lurie Cancer Center, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - University of Iowa, Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Michigan State University, Breslin Cancer Center, Lansing, Michigan
  - University of Minnesota: Masonic Cancer Center, Minneapolis, Minnesota
  - University of Nebraska, Fred and Pamela Buffet Cancer Center, Omaha, Nebraska
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Penn State Hershey Cancer Institute, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dudek AZ, Liu LC, Gupta S, Logan TF, Singer EA, Joshi M, Zakharia YN, Lang JM, Schwarz JK, Al-Janadi A, Alva AS. Phase Ib/II Clinical Trial of Pembrolizumab With Bevacizumab for Metastatic Renal Cell Carcinoma: BTCRC-GU14-003. J Clin Oncol. 2020 Apr 10;38(11):1138-1145. doi: 10.1200/JCO.19.02394. Epub 2020 Feb 25. PMID 32097091
- See also: Big Ten Cancer Research Consortium Website — http://www.bigtencrc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A - Phase 1b Dose Escalation Cohort: Cohort 1 will consist of 3-6 patients who will receive MK-3475 200mg and bevacizumab 10mg on day 1 of the 21-day cycle. The drugs are administered 15-30 minutes apart in separate intravenous infusions.
  If none of the 3 subjects experience a dose limiting toxicity (DLT) during the first cycle of therapy, an additional 3 subjects will be enrolled at dose level 2. If all three subjects in dose level 2 complete the first cycle of therapy without DLT, 3 more subjects will be enrolled to ensure only 0-1 of 6 subjects have a DLT. There will be no further escalation beyond dose level 2.
  MK-3475: Arm A: Phase 1b Cohort 1: 200mg IV; Arm A: Phase 1b Cohort 2: 200mg IV
  Bevacizumab: Arm A: Phase 1b Cohort 1: 10mg IV;
- Arm A - Phase Ib Dose Ecalation Cohort 2: Cohort 2 will consist of 3-9 patients who will receive MK-3475 200mg and bevacizumab 15mg on day 1 of the 21-day cycle. The drugs are administered 15-30 minutes apart in separate intravenous infusions.
  If none of the 3 subjects experience a dose limiting toxicity (DLT) during the first cycle of therapy, an additional 3 subjects will be enrolled at dose level 2. If all three subjects in dose level 2 complete the first cycle of therapy without DLT, 3 more subjects will be enrolled to ensure only 0-1 of 6 subjects have a DLT. There will be no further escalation beyond dose level 2.
  MK-3475: Arm A: Phase 1b Cohort 1: 200mg IV; Arm A: Phase 1b Cohort 2: 200mg IV
  Bevacizumab: Arm A: Phase 1b Cohort 2: 15mg IV
- Arm B - Phase II Investigational Treatment: The maximum safe dose of MK-3475 in combination bevacizumab (as determined in the phase 1b cohort) will be given on day 1 of each 21 day cycle.
  MK-3475: Arm B: Phase II Treatment: 200mg IV
  Bevacizumab: Arm B: Phase II Treatment: administered at the maximum safe dose of 5mg or 10mg as established in the Phase 1b dose escalation cohort study.
Period: Overall Study
Arm/Group | Arm A - Phase 1b Dose Escalation Cohort | Arm A - Phase Ib Dose Ecalation Cohort 2 | Arm B - Phase II Investigational Treatment
Started | 3 | 10 | 48
Completed | 0 | 0 | 29
Not Completed | 3 | 10 | 19
Not completed — Adverse Event | 2 | 3 | 3
Not completed — Disease Progression | 1 | 5 | 16
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Symptomatic Deterioration | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: No per-group analysis was completed in the dose escalation cohort because the Phase IB dose-finding study found no dose-limiting toxicities and the primary objective (determine MTD) was satisfied. The baseline demographics as presented have been presented in several abstracts and published in the Journal of Clinical Oncology.
Groups:
- Arm A - Phase 1b Dose Escalation Cohort: Cohort 1 will consist of 3-6 patients who will receive MK-3475 200mg and bevacizumab 10mg on day 1 of the 21-day cycle. The drugs are administered 15-30 minutes apart in separate intravenous infusions.
  Cohort 2 will consist of 3-9 patients who will receive MK-3475 200mg and bevacizumab 15mg on day 1 of the 21-day cycle. The drugs are administered 15-30 minutes apart in separate intravenous infusions.
  If none of the 3 subjects experience a dose limiting toxicity (DLT) during the first cycle of therapy, an additional 3 subjects will be enrolled at dose level 2. If all three subjects in dose level 2 complete the first cycle of therapy without DLT, 3 more subjects will be enrolled to ensure only 0-1 of 6 subjects have a DLT. There will be no further escalation beyond dose level 2.
  MK-3475: Arm A: Phase 1b Cohort 1: 200mg IV; Arm A: Phase 1b Cohort 2: 200mg IV
  Bevacizumab: Arm A: Phase 1b Cohort 1: 10mg IV; Arm A: Phase 1b Cohort 2: 15mg IV
- Total: Total of all reporting groups
Arm/Group | Arm A - Phase 1b Dose Escalation Cohort | Arm B - Phase II Investigational Treatment | Total
Number analyzed (Participants) | 13 | 48 | 61
Age, Continuous [Median (Full Range); unit: years] | 55 [33 to 68] | 61 [42 to 84] | 60 [33 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 15 | 17
  Male | 11 | 33 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 5
  Not Hispanic or Latino | 10 | 38 | 48
  Unknown or Not Reported | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 45 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 13 | 48 | 61
Karnofsky Performance Status (KPS) [Count of Participants; unit: Participants] — KPS is a general indicator of a subject's well being and ability to carry on daily activities.
  100:Normal no complaints 90:Able to carry on normal activity 80:Normal activity with effort; some signs or symptoms of disease. 70:Cares for self 60:Requires occasional assistance, but is able to care for most of his personal needs. 50:Requires considerable assistance and frequent medical care.
  40:Disabled 30:Severely disabled 20:Very sick 10:Moribund 0:Dead
  Participants
    KPS 70 | 2 | 3 | 5
    KPS 80 | 3 | 10 | 13
    KPS 90 | 1 | 20 | 21
    KPS 100 | 7 | 15 | 22
Prior Nephrectomy [Count of Participants; unit: Participants]
  Yes | 11 | 43 | 54
  No | 2 | 5 | 7
Bone Metastases [Count of Participants; unit: Participants]
  Yes | 6 | 10 | 16
  No | 7 | 38 | 45
Metastatic RCC Prognosis (by IMDC/Heng Score) [Count of Participants; unit: Participants] — The IMDC\Heng Score is calculated based on the number of risk factors:
  0 Risk Factors: Favorable Prognosis 1-2 Risk Factors: Intermediate Prognosis 3-6 Risk Factors: Poor Prognosis
  Participants
    Favorable | 5 | 10 | 15
    Intermediate | 3 | 31 | 34
    Poor | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Maximum Safe Dose of Treatment Regimen
Description: To establish the maximum tested safe dose of bevacizumab in combination with 200mg of MK-3475(pembrolizumab) for subjects with metastatic clear cell renal carcinoma after failure of at least one systemic therapy for metastatic disease.
Time Frame: Every 21 days while on treatment (estimated 4 months)
Measure: Number; unit: mg/kg
Arm/Group | Arm A - Phase 1b Dose Escalation Cohort
Number analyzed (Participants) | 13
mg/kg | 15

2. Primary Outcome: Overall Response Rate
Description: To determine the activity of combination of MK-3475 and bevacizumab in first line therapy for subjects with treatment naïve metastatic clear cell RCC as assessed by response rates (complete or partial response) By calculating the proportion of subjects with a response (CR, PR) based on RECIST 1.1 where:
  Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started
Time Frame: Every 6 weeks while on treatment (estimated 10 months)
Population: Results for Arm A - Phase Ib are reported as a single group, no per-group analyses were planned or performed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A - Phase 1b Dose Escalation Cohort | Arm B - Phase II Investigational Treatment
Number analyzed (Participants) | 13 | 48
percentage of participants | 41.7 [15.2 to 72.3] | 60.9 [45.4 to 74.9]

3. Secondary Outcome: Progression-Free Survival
Description: To determine median progression-free survival (PFS) for this patient population, per RECIST 1.1 where:
  Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started
Time Frame: Up to two years from enrollment
Population: Results for Arm A - Phase Ib are reported as a single group, no per-group analyses were planned or performed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A - Phase 1b Dose Escalation Cohort | Arm B - Phase II Investigational Treatment
Number analyzed (Participants) | 13 | 47
months | 9.9 [4.9 to 16.7] | 20.7 [11.3 to 27.4]

4. Secondary Outcome: Overall Survival
Description: To determine if treatment regimen improves overall survival for this patient population. Median overall survival will be calculated up to 2 years from registration.
Time Frame: Up to 2 years from registration
Population: Results for Arm A - Phase Ib are reported as a single group, no per-group analyses were planned or performed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Phase 1b Dose Escalation Cohort | Arm B - Phase II Investigational Treatment
Number analyzed (Participants) | 13 | 47
Months | 17.9 [6.3 to NA] — 95% confidence interval upper limit not estimable | NA [NA to NA] — Median OS was not reached (only 15 of 47 evaluable subjects died)

5. Secondary Outcome: Clinical Benefit Rate
Description: To determine the proportion of subjects with clinical benefit (complete response, partial response, or stable disease) based on RECIST 1.1, where:
  Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started
Time Frame: Every 6 months while on treatment (estimated 4-10 months)
Population: Results for Arm A - Phase Ib are reported as a single group, no per-group analyses were planned or performed.
Measure: Number; unit: percentage of subjects
Arm/Group | Arm A - Phase 1b Dose Escalation Cohort | Arm B - Phase II Investigational Treatment
Number analyzed (Participants) | 13 | 46
percentage of subjects | 91.67 | 100

6. Secondary Outcome: Characterize Adverse Events
Description: Characterize adverse effects (AE) of pembrolizumab in combination with bevacizumab in subjects with metastatic RCC after failure of at least one systemic therapy. Toxicity will be assessed using CTCAE version 4. All grade 3 and 4 treatment-related adverse events will be reported.
Time Frame: Every week while on treatment (estimated 4-10 months)
Population: The analysis population for this objective was defined in the protocol as "all subjects who received at least one dose of study drug". No per-arm or per-cohort analyses were planned or performed.
Measure: Number; unit: events
Groups:
- All Subjects: Adverse events are summarized for all study participants who received at least one dose of study drug.
Arm/Group | All Subjects
Number analyzed (Participants) | 60
events
  Duodenal ulcer: Grade 4 | 1
  Hyponatremia: Grade 4 | 1
  Hypertension: Grade 3 | 15
  Proteinuria: Grade 3 | 6
  Adrenal insufficiency: Grade 3 | 4
  Pain/Headaches: Grade 3 | 3
  Pneumonitis: Grade 3 | 2
  Hyponatremia: Grade 3 | 2
  Generalized muscle weakness: Grade 3 | 2
  Dehydration: Grade 3 | 2
  Skin Rashes: Grade 3 | 2
  Anemia: Grade 3 | 2
  Nausea: Grade 3 | 1
  Vomiting: Grade 3 | 1
  Thromboembolic event: Grade 3 | 1
  Seizure: Grade 3 | 1
  Myocardial infarction: Grade 3 | 1
  Mucositis oral: Grade 3 | 1
  Immune mediated hepatitis: Grade 3 | 1
  Immune mediated gastritis: Grade 3 | 1
  Hypothyroidism | 1
  Hematuria | 1
  Flu like symptoms: Grade 3 | 1
  Diarrhea: Grade 3 | 1
  Arthralgia: Grade 3 | 1
  Alkaline phosphatase increased: Grade 3 | 1

ADVERSE EVENTS:
Time Frame: Every week while on treatment (estimated 4-10 months)
Groups:
- All Subjects: Adverse events are summarized for all study participants who received at least one dose of study drug. Per the protocol, the safety analysis population "will comprise all subjects who received at least one dose of study drug". Consequently, no per-group analyses were planned or performed.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 28/61
Serious Adverse Events (participants affected / at risk) | 32/61
Other Adverse Events (participants affected / at risk) | 60/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=61)
ABDOMINAL INFECTION (Infections and infestations) | 1 (1)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 (2)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 5 (5)
ANEMIA (Blood and lymphatic system disorders) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
BUTTOCK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
CARDIAC DISORDERS (Cardiac disorders) | 1 (1)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1)
DUODENAL ULCER (Gastrointestinal disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 2 (2)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
HEART FAILURE (Cardiac disorders) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 1 (2)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1)
INFECTIONS AND INFESTATIONS (Infections and infestations) | 1 (1)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1)
PAIN (General disorders) | 2 (2)
PANCREATITIS (Gastrointestinal disorders) | 1 (1)
PELVIC PAIN (Reproductive system and breast disorders) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 3 (3)
PROTEINURIA (Renal and urinary disorders) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (2)
SMALL INTESTINE INFECTION (Infections and infestations) | 1 (1)
SOFT TISSUE INFECTION (Infections and infestations) | 1 (1)
STROKE (Nervous system disorders) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1)
TRANSIENT ISCHEMIC ATTACKS (Nervous system disorders) | 1 (1)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
VASCULAR DISORDERS (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=61)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 10 (15)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 5 (6)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 3 (3)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 3 (5)
ADULT RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 9 (15)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 11 (16)
ALLERGIC REACTION (Immune system disorders) | 2 (2)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 3 (3)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1)
ANAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 12 (18)
ANOREXIA (Metabolism and nutrition disorders) | 25 (35)
ANXIETY (Psychiatric disorders) | 6 (7)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7 (10)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 10 (10)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 12 (17)
ATAXIA (Nervous system disorders) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 16 (21)
BLOATING (Gastrointestinal disorders) | 2 (2)
BLOOD AND LYMPHATIC SYSTEM DISORDERS (Blood and lymphatic system disorders) | 2 (3)
BLOOD BILIRUBIN INCREASED (Investigations) | 5 (8)
BLURRED VISION (Eye disorders) | 3 (3)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 5 (5)
BREAST PAIN (Reproductive system and breast disorders) | 1 (1)
BRONCHIAL INFECTION (Infections and infestations) | 1 (1)
BRUISING (Injury, poisoning and procedural complications) | 4 (4)
BURN (Injury, poisoning and procedural complications) | 2 (2)
BUTTOCK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
CARDIAC DISORDERS (Cardiac disorders) | 4 (4)
CHEST PAIN - CARDIAC (Cardiac disorders) | 1 (1)
CHILLS (General disorders) | 5 (5)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1)
CHOLESTEROL HIGH (Investigations) | 5 (5)
COGNITIVE DISTURBANCE (Nervous system disorders) | 1 (1)
COLITIS (Gastrointestinal disorders) | 2 (4)
CONSTIPATION (Gastrointestinal disorders) | 25 (34)
COUGH (Respiratory, thoracic and mediastinal disorders) | 25 (34)
CREATININE INCREASED (Investigations) | 21 (38)
DEHYDRATION (Metabolism and nutrition disorders) | 6 (9)
DENTAL CARIES (Gastrointestinal disorders) | 2 (2)
DEPRESSION (Psychiatric disorders) | 6 (7)
DIARRHEA (Gastrointestinal disorders) | 25 (40)
DIZZINESS (Nervous system disorders) | 12 (15)
DRY EYE (Eye disorders) | 2 (3)
DRY MOUTH (Gastrointestinal disorders) | 4 (4)
DRY SKIN (Skin and subcutaneous tissue disorders) | 10 (12)
DYSGEUSIA (Nervous system disorders) | 7 (7)
DYSPEPSIA (Gastrointestinal disorders) | 5 (5)
DYSPHAGIA (Gastrointestinal disorders) | 4 (4)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 12 (17)
EAR AND LABYRINTH DISORDERS (Ear and labyrinth disorders) | 1 (1)
EAR PAIN (Ear and labyrinth disorders) | 1 (1)
EDEMA FACE (General disorders) | 1 (1)
EDEMA LIMBS (General disorders) | 19 (24)
ENDOCRINE DISORDERS (Endocrine disorders) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 10 (14)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 1 (1)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 1 (1)
EYE DISORDERS (Eye disorders) | 4 (6)
EYE PAIN (Eye disorders) | 2 (2)
FALL (Injury, poisoning and procedural complications) | 5 (5)
FATIGUE (General disorders) | 44 (66)
FEVER (General disorders) | 3 (3)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 3 (4)
FLATULENCE (Gastrointestinal disorders) | 3 (3)
FLU LIKE SYMPTOMS (General disorders) | 3 (4)
FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 3 (3)
GASTRITIS (Gastrointestinal disorders) | 4 (5)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 8 (9)
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 13 (18)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS (General disorders) | 8 (15)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 5 (5)
GENITAL EDEMA (Reproductive system and breast disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 25 (34)
HEMATURIA (Renal and urinary disorders) | 9 (13)
HEMOGLOBIN INCREASED (Investigations) | 2 (5)
HEMORRHOIDAL HEMORRHAGE (Gastrointestinal disorders) | 2 (2)
HEMORRHOIDS (Gastrointestinal disorders) | 3 (3)
HEPATOBILIARY DISORDERS (Hepatobiliary disorders) | 2 (2)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 8 (8)
HOT FLASHES (Vascular disorders) | 1 (1)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 10 (13)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 11 (22)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 2 (2)
HYPERKALEMIA (Metabolism and nutrition disorders) | 15 (19)
HYPERNATREMIA (Metabolism and nutrition disorders) | 3 (3)
HYPERPARATHYROIDISM (Endocrine disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 39 (93)
HYPERTHYROIDISM (Endocrine disorders) | 3 (3)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 8 (10)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 4 (4)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 4 (4)
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPONATREMIA (Metabolism and nutrition disorders) | 11 (27)
HYPOTENSION (Vascular disorders) | 5 (5)
HYPOTHYROIDISM (Endocrine disorders) | 14 (16)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 3 (3)
INFECTIONS AND INFESTATIONS (Infections and infestations) | 4 (4)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS (Injury, poisoning and procedural complications) | 3 (3)
INR INCREASED (Investigations) | 2 (2)
INSOMNIA (Psychiatric disorders) | 12 (14)
INVESTIGATIONS (Investigations) | 10 (20)
IRRITABILITY (General disorders) | 1 (1)
LEFT VENTRICULAR SYSTOLIC DYSFUNCTION (Cardiac disorders) | 1 (1)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 3 (4)
LIP INFECTION (Infections and infestations) | 1 (1)
LIPASE INCREASED (Investigations) | 1 (1)
LOCALIZED EDEMA (General disorders) | 3 (3)
LOWER GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1)
LUNG INFECTION (Infections and infestations) | 1 (1)
LYMPHEDEMA (Vascular disorders) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 2 (2)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1)
MENOPAUSE (Social circumstances) | 1 (1)
METABOLISM AND NUTRITION DISORDERS (Metabolism and nutrition disorders) | 2 (2)
MUCOSITIS ORAL (Gastrointestinal disorders) | 9 (14)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER (Musculoskeletal and connective tissue disorders) | 22 (29)
MYALGIA (Musculoskeletal and connective tissue disorders) | 7 (8)
NAIL INFECTION (Infections and infestations) | 1 (1)
NAIL RIDGING (Skin and subcutaneous tissue disorders) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 27 (38)
NECK EDEMA (General disorders) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
NERVOUS SYSTEM DISORDERS (Nervous system disorders) | 5 (5)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 2 (2)
ORAL DYSESTHESIA (Gastrointestinal disorders) | 4 (4)
ORAL PAIN (Gastrointestinal disorders) | 2 (2)
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 1 (2)
PAIN (General disorders) | 12 (14)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 16 (28)
PALMAR-PLANTAR ERYTHRODYSESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 3 (3)
PALPITATIONS (Cardiac disorders) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 2 (2)
PAPULOPUSTULAR RASH (Infections and infestations) | 1 (1)
PARESTHESIA (Nervous system disorders) | 1 (1)
PERIORBITAL EDEMA (Skin and subcutaneous tissue disorders) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2 (2)
PLATELET COUNT DECREASED (Investigations) | 6 (9)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 4 (5)
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 6 (8)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 7 (8)
PROTEINURIA (Renal and urinary disorders) | 24 (62)
PRURITUS (Skin and subcutaneous tissue disorders) | 20 (24)
PSYCHIATRIC DISORDERS (Psychiatric disorders) | 1 (1)
PURPURA (Skin and subcutaneous tissue disorders) | 1 (1)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 19 (27)
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1)
RENAL AND URINARY DISORDERS (Renal and urinary disorders) | 10 (15)
REPRODUCTIVE SYSTEM AND BREAST DISORDERS (Reproductive system and breast disorders) | 2 (2)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS (Respiratory, thoracic and mediastinal disorders) | 13 (20)
RHINITIS INFECTIVE (Infections and infestations) | 1 (2)
SEIZURE (Nervous system disorders) | 2 (3)
SERUM AMYLASE INCREASED (Investigations) | 1 (1)
SINUS BRADYCARDIA (Cardiac disorders) | 4 (4)
SINUS PAIN (Nervous system disorders) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 2 (2)
SINUSITIS (Infections and infestations) | 7 (12)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS (Skin and subcutaneous tissue disorders) | 22 (32)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 2 (2)
SKIN INFECTION (Infections and infestations) | 3 (3)
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 1 (1)
SLEEP APNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 2 (2)
SOFT TISSUE INFECTION (Infections and infestations) | 1 (2)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 2 (2)
STOMACH PAIN (Gastrointestinal disorders) | 3 (3)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1)
SURGICAL AND MEDICAL PROCEDURES (Surgical and medical procedures) | 3 (4)
TESTICULAR DISORDER (Reproductive system and breast disorders) | 1 (1)
TESTICULAR PAIN (Reproductive system and breast disorders) | 4 (4)
THROMBOEMBOLIC EVENT (Vascular disorders) | 2 (3)
TOOTH INFECTION (Infections and infestations) | 3 (5)
TOOTHACHE (Gastrointestinal disorders) | 2 (2)
TREMOR (Nervous system disorders) | 2 (2)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 15 (22)
URINARY FREQUENCY (Renal and urinary disorders) | 2 (3)
URINARY INCONTINENCE (Renal and urinary disorders) | 1 (2)
URINARY RETENTION (Renal and urinary disorders) | 3 (3)
URINARY TRACT INFECTION (Infections and infestations) | 8 (9)
URINARY TRACT PAIN (Renal and urinary disorders) | 1 (1)
URINARY URGENCY (Renal and urinary disorders) | 1 (1)
VASCULAR DISORDERS (Vascular disorders) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1)
VOICE ALTERATION (Respiratory, thoracic and mediastinal disorders) | 4 (4)
VOMITING (Gastrointestinal disorders) | 15 (27)
WATERING EYES (Eye disorders) | 3 (3)
WEIGHT GAIN (Investigations) | 8 (9)
WEIGHT LOSS (Investigations) | 18 (19)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-11): https://cdn.clinicaltrials.gov/large-docs/08/NCT02348008/Prot_SAP_000.pdf